CLINICAL TRIAL: NCT00756808
Title: Is Tuberculin Skin Testing Effective in Screening for Latent TB in Elderly Residents of Nursing Homes? Comparison With a New IFN-y Based Assay
Brief Title: Is Tuberculin Skin Testing Effective in Screening for Latent Tuberculosis (TB) in Elderly Residents of Nursing Homes?
Status: Completed | Type: Observational
Sponsor: Northwell Health (Other)
Collaborators: Staten Island University Hospital (Other)
Responsible Party: Principal Investigator, Donna Seminara, Program Director, Geriatric Medicine, Northwell Health
Other Study IDs: 07-050
Record Dates: First submitted 2008-09-19; First posted 2008-09-22 (Estimated); Last update posted 2014-02-07 (Estimated); Status verified 2014-02

CONDITIONS: Tuberculosis
Keywords: latent tuberculosis in elderly
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
In face of the increased rates of tuberculosis in residents of long term care facilities, annual screening for latent tuberculosis is recommended. Tuberculin skin testing using purified protein derivative (PPD) is used for this purpose. Sensitivity of the PPD testing is, however, dependent on a normal T cell function. It is now evident that the immune system undergoes age-associated alteration known as immune senescence. The depressed T-cell responses may clinically manifest as attenuated delayed-type hypersensitivity. This attenuated reaction may affect the sensitivity of the PPD in detection of latent TB in the elderly.

This prospective study will examine the utility of interferon-gamma (IFN-γ) based assay, T-SPOT.TB, for detection of latent tuberculosis in nursing home patients who are 65 years of age or older.

ELIGIBILITY:
Inclusion Criteria:

* 65 years of age and older
* No ulcerating or blistering skin disorder
* No previous history of adverse reaction to PPD testing
* No blood transfusion within 6 weeks prior to enrollment
* If the participant had a PPD placed and read by a public health department representative within the last 6 months, repeat PPD will not be done, but the person may participate in the study
* Participant may have been Bacille de Calmette et Guerin (BCG)-vaccinated

Exclusion Criteria:

* Less than 65 years
* Not a resident of a long term care facility
* Diagnosis of Tuberculosis
* blood transfusion within 6 weeks of enrollment
* Prior diagnosis of immune deficiency

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: 65 and older
Sampling Method: Non-Probability Sample
Enrollment: 135 (Actual)
Dates: Start 2007-10; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
detection of latent TB | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Donna Seminara, MD, Principal Investigator — Staten Island University Hospital
Locations (1):
- Staten Island University Hospital, Staten Island, New York, United States